CLINICAL TRIAL: NCT00957190
Title: Change in Optic Nerve Head Blood Flow,Optic Nerve Topography and Diurnal Fluctuation of Intraocular Pressure and Pulsatile Ocular Blood Flow in Glaucoma:Cosopt and Xalatan vs Xalatan Alone
Brief Title: The DIOXXACT Trial(Diurnal IOP and OBF Xalatan vs Xalatan And Cosopt Trial)
Acronym: DIOXXACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mark R. Lesk, Director of opthalmology research, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 157-00; IISP34708 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2009-08-04; First posted 2009-08-12 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Eye Disease
Keywords: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Eye Diseases; Ocular Hypertension; Glaucoma, Open-Angle | interventions — dorzolamide; Timolol; dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cosopt (Experimental): Cosopt ('Dorzolamide 20 mg and Timolol 5 mg) bid And Xalatan hs Vs Xalatan hs Alone
  Interventions: Drug: Dorzolamide 20 mg and Timolol 5 mg

INTERVENTIONS:
Drug: Dorzolamide 20 mg and Timolol 5 mg — Twice daily in the affected eye(s)
  Other Names: Cosopt

SUMMARY:
Diurnal and intervisit fluctuations in IOP are strongly associated with progression of open angle glaucoma and therefore need to be minimized. Control of diurnal fluctuations of IOP with different ocular hypotensive medications has been studied in some detail. But how do IOP changes contribute to progressive glaucomatous optic nerve damage? It is reasonable to assume that there are two principal effects of IOP changes. First, IOP fluctuations result in changes in the stresses and strains on the ONH which in turn result in morphological changes to the ONH. These morphological changes could in turn result in stretching and damage to axons of the ONH. Secondly, IOP fluctuations results in changes to the forces acting on the ONH vasculature, leading to changes in ONH vascular perfusion. These changes to perfusion could in turn result in relative ischemia of the ONH and consequent ONH damage.

The investigators propose to monitor diurnal fluctuations in IOP and choroidal blood flow (Pulsatile Ocular Blood Flow,POBF), and intervisit ONH topographical and blood flow changes-ie to monitor the direct ONH consequences of IOP . Open angle glaucoma patients are commonly prescribed topical latanoprost as first line therapy. The EXACCT study, for which I was the principal investigator and which is now submitted for publication, demonstrated that COSOPT was an efficacious choice as second line therapy for patients not controlled on latanoprost monotherapy. The investigators will therefore recruit 20 OAG patients on latanoprost monotherapy, perform diurnal curves of IOP, as well as a.m. ONH morphology and ONH blood flow. Cosopt will then be added and at the next visit the same measurements will be repeated.

The investigators expect that when Cosopt is added the investigators will demonstrate improved IOP, morphology and blood flow compared to the latanoprost baseline. Furthermore the investigators expect the the diurnal fluctuation of IOP and choroidal blood flow will be stabilized on Cosopt therapy. The implications are that adding Cosopt to latanoprost can stabilize not only the IOP but also the damaging consequences of IOP to the optic nerve head.

DETAILED DESCRIPTION:
Twenty patients with open angle glaucoma or ocular hypertension currently on latanoprost immunotherapy will be recruited.

A complete routine ophthalmic examination including biomicroscopy, gonioscopy and fundus ophthalmoscopy will be performed. The eye with better visual acuity is selected for fundus flowmetry.

All patients will undergo a complete diurnal workup including IOP, as well as 10am Confocal scanning laser ophthalmoscopy (Heidelberg Retina Tomography-3) of ONH topography. Optic nerve head, nasal and temporal peripapillary retinal blood flow are measured with scanning laser Doppler flowmetry (SLDF; Heidelberg Retinal Flowmeter/Tomograph, SLDF analysis software v3.3, Heidelberg Engineering, Germany Goldmann IOP will be measured at 8am, 10am 2pm and 4pm. Pulse amplitude, similar to Pulsatility Ocular Blood Flow (POBF) will be measured using the Pascal Dynamic Contour Tonometer (DCT) at 8am, 10am, 2pm, and 4 pm.

All procedures will conform to the Declaration of Helsinki and the study will be approved by the Ethics Committee and each patient will sign an informed consent form.

Following visit one, Cosopt will be added to the patients therapy (bid). Following 6 weeks of therapy patients will return for visit two. Cosopt will be applied by the investigator at 8am on visit 2.

We expect that this blood flow will be improved with COSOPT therapy and that the diurnal fluctuation of this parameter will be improved as well. It is evidently of great interest to examine diurnal changes in ocular blood flow with and without COSOPT and the measurement of POBF can be performed without great cost and is well tolerated by the patient.

Changes in IOP, ONH Topography, and ONH blood flow will be analysed using appropriate statistical approaches

ELIGIBILITY:
Inclusion Criteria:

* Subjets with open angle glaucoma or ocular hypertension currently on latanoprost immunotherapy.
* Subjets must have clear media, corrected visual acuity of 6/12 or better,and be able to sit for imaging.

Exclusion Criteria:

* Subjets with contraindications or known allergies to any of the components of Cosopt.
* Subjets who had undergoing laser or any ocular surgery.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-05-04 (Actual); Primary Completion 2011-09-14 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Clinical evidence for lower diurnal variational Intraocular Pressure | Six weeks

SECONDARY OUTCOMES:
The Intraocular Pressure, Retinal and choroidal blood flow will be stabilized on Cosopt therapy | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Lesk, MSc,MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hafez AS, Bizzarro RL, Rivard M, Trabut I, Lovasik JV, Kergoat H, Lesk MR. Reproducibility of retinal and optic nerve head perfusion measurements using scanning laser Doppler flowmetry. Ophthalmic Surg Lasers Imaging. 2003 Sep-Oct;34(5):422-32. PMID 14509472
- [Result] Yoshida A, Feke GT, Mori F, Nagaoka T, Fujio N, Ogasawara H, Konno S, Mcmeel JW. Reproducibility and clinical application of a newly developed stabilized retinal laser Doppler instrument. Am J Ophthalmol. 2003 Mar;135(3):356-61. doi: 10.1016/s0002-9394(02)01949-9. PMID 12614754
- [Result] Lesk MR, Hafez AS, Descovich D. Relationship between central corneal thickness and changes of optic nerve head topography and blood flow after intraocular pressure reduction in open-angle glaucoma and ocular hypertension. Arch Ophthalmol. 2006 Nov;124(11):1568-72. doi: 10.1001/archopht.124.11.1568. PMID 17102003
- [Result] Michelson G, Schmauss B. Two dimensional mapping of the perfusion of the retina and optic nerve head. Br J Ophthalmol. 1995 Dec;79(12):1126-32. doi: 10.1136/bjo.79.12.1126. PMID 8562550
- [Result] Sehi M, Flanagan JG, Zeng L, Cook RJ, Trope GE. Anterior optic nerve capillary blood flow response to diurnal variation of mean ocular perfusion pressure in early untreated primary open-angle glaucoma. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4581-7. doi: 10.1167/iovs.05-0209. PMID 16303952